CLINICAL TRIAL: NCT02567513
Title: Cost-Effectiveness of Weight Loss Prevention in Nursing Homes: A Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sandra Simmons, Associate Professor of Medicine, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 090948
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Weight Loss
Keywords: food and fluid intake; nursing homes
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care control group (No Intervention): Eligible, consented residents continue to receive usual care from nursing home staff and are independently monitored by trained research staff.
- Supplement Intervention (Experimental): Residents are offered a variety of supplement types and flavors consistent with prescribed orders twice per day (morning and afternoon), five days per week, for 24 consecutive weeks by trained research personnel. Research staff also provide the appropriate level and amount of assistance to encourage consumption.
  Interventions: Behavioral: Supplement Intervention
- Snack Intervention (Experimental): Residents are offered a variety of snack options (foods and fluids, including supplement) consistent with prescribed orders twice per day (morning and afternoon), five days per week, for 24 consecutive weeks by trained research personnel. Research staff also provide the appropriate level and amount of assistance to encourage consumption.
  Interventions: Behavioral: Snack Intervention

INTERVENTIONS:
Behavioral: Supplement Intervention — Supplements given twice/day, 5 days/week, for 24 weeks by research staff.
  Other Names: Experimental Supplement Intervention
  Arms: Supplement Intervention
Behavioral: Snack Intervention — Snacks given twice/day, 5 days/week for 24 weeks by research staff.
  Other Names: Experimental Snack Intervention
  Arms: Snack Intervention

SUMMARY:
Low oral food and fluid intake and unintentional weight loss are common problems among long-stay nursing home (NH) residents and are associated with adverse, costly clinical outcomes. This study will use a controlled, intervention design to determine the cost-effectiveness of oral liquid nutrition supplements with an alternative nutrition intervention that offers NH residents a choice between supplements and other foods and fluids (i.e., snacks) between meals in a group of 200 residents across 4 NH sites. Residents with an order for supplementation will be included in this study and randomized into one of three groups: (1) usual care control; (2) oral liquid nutrition supplementation intervention; or (3) choice intervention. The usual care control group will continue to receive standard NH care for supplement or snack delivery. Research staff will provide the same supplements used by the NH (group two) or a choice between supplements and other foods and fluids (group three) twice daily, five days per week, for 24 weeks and document the daily costs of intervention implementation when also providing a prompting protocol known to improve intake and enhance independence in eating. Based on extensive preliminary data, it is anticipated that both groups two and three will require significantly more staff time than usual care (group one). Thus, the labor costs of these interventions will be documented and compared to effectiveness measures. Effectiveness measures include the following resident outcomes: improvements in total daily caloric intake, weight, nutrition and hydration status and quality of life. These outcomes will be independently monitored for all three groups across 24-weeks by trained research staff using standardized, validated protocols.

ELIGIBILITY:
Inclusion Criteria:

* Long-stay nursing home residents,
* capable of oral food and fluid intake,
* physician or dietitian order for caloric supplementation.

Exclusion Criteria:

* Short-stay nursing home residents (rehabilitation),
* feeding tube,
* hospice care.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Total caloric intake during and between meals | 24 weeks
  Weighed intake methods both during and between meals were used to assess total caloric intake before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra F Simmons, PhD, Principal Investigator — Vanderbilt University